CLINICAL TRIAL: NCT01452477
Title: Effect of Tanshinone on Hormonal and Metabolic Features in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Tanshinone in Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Chairman Dept Obs & Gyn, First Affiliated Hospital, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tanshinone-HLJUCM
Record Dates: First submitted 2011-10-06; First posted 2011-10-14 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Cryptotanshinone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — tanshinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tanshinone (Active Comparator): tanshinone 1.0g / time, 3 times / day orally, continuous treatment for 12 weeks.
  Interventions: Drug: tanshinone
- tanshinone placebo (Placebo Comparator): placebo 1.0g / time, 3 times / day orally, continuous treatment for 12 weeks.
  Interventions: Drug: tanshinone placebo

INTERVENTIONS:
Drug: tanshinone — tanshinone 1.0g / time, 3 times / day orally, continuous treatment for 12 weeks.
  Arms: tanshinone
Drug: tanshinone placebo — placebo 1.0g / time, 3 times / day orally, continuous treatment for 12 weeks.
  Arms: tanshinone placebo

SUMMARY:
Tanshinone was originally isolated from dried roots of Salvia miltiorrhiza bunge. In Chinese medicine, this herb has been widely prescribed for several pathologies, including diabetes, acne, cardiovascular disease.It has been demonstrated that the therapeutic benefit of cryptotanshinone on prenatally androgenized rats may be mediated by its dual regulation of key molecules during both insulin signaling and androgen synthesis.The purpose of this study is to determine whether tanshinone may prove effective in eradicating Polycystic Ovary Syndrome (PCOS) symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Presence of PCOS diagnosed based on the Androgen Excess Society criteria. All subjects must have hyperandrogenism (hirsutism and/or hyperandrogenemia), ovarian dysfunction (oligoanovulation and/or polycystic ovaries), and exclusion of other androgen excess related disorders. Oligomenorrhea is defined as an intermenstrual interval >35 days or <8 menstrual bleedings in the past year. Amenorrhea is defined as an intermenstrual interval >90 days. Clinical hyperandrogenism is defined as a Ferriman-Gallwey (FG) score ≥5
* Age of women from 18 to 35 years；
* No desire of children within 6 month and use condoms for contraception.

Exclusion Criteria:

* Use of hormonal drugs or other medications, which can affect the results of the study especially Chinese herbal prescriptions in the past 12 weeks；
* Patients with other androgen excess endocrine disorders including 21-hydroxylase deficiency, hyperprolactinemia, Cushing syndrome, severe insulin resistance, thyroid dysfunction；
* Patients with history of sever cardiac , pulmonary, hepatic, renal, neurologic disease or mental illness；
* Pregnancy or lactation.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
basal testosterone | 3 months
  The primary outcome measure is a decrease in basal testosterone.

SECONDARY OUTCOMES:
Ovarian androgen biosynthesis | 3 months
  Human chorionic gonadotropin (HCG) induced response of androgens including 17-hydroxyprogesterone (17-OHP), androstenedione (A2), testosterone (T)
Whole body insulin action | 3 months
  Insulin resistance by the glucose disposal rate (GDR) with hyperinsulinemic euglycemic clamp test
Oral glucose tolerance test (OGTT) | 3 months
  All the participants will undergo an overnight fast. After ingestion of a 75-g glucose load, blood samples will be obtained at 0, 30, 60, 90, and 120min for glucose and insulin level determination.
Reproductive hormones | 3 months
  estradiol (E2), 17-α-hydroxyprogesterone (17-OHP), follicle stimulation hormone (FSH), leutinizing hormone (LH), sex hormone binding globulin and dehydroepiandrosterone sulphate.
Fasting gluco-lipid metabolic profiles | 3 months
quality of life | 3 months
  the quality of life will be assessed by the Polycystic Ovary Syndrome Questionnaire (PCOS-QOL)and the Chinese Quality of Life (ChQOL).
Weight, waist/hip circumference, blood pressure, F-G score and acne before and after treatment | 3 months
Adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoke Wu, docotor, Study Chair — The First Affliated Hospital,Heilongjiang University of Chinese Medicine .
Locations (4):
- China (4):
  - Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Huaian Maternal and Child Health Hospital, Huaian, Jiangsu
  - Lianyungang Maternal and Child Health Hospital, Lianyungang, Jiangsu
  - JiangXi University of Traditional Chinese Medicine, Nanchang, Jiangxi